CLINICAL TRIAL: NCT03367273
Title: Study of the Cutaneous Expression of Thymic Stromal Lymphopoietin (TSLP) in a Sample of Vitiligo Patients
Brief Title: Thymic Stromal Lymphopoietin (TSLP) in Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, Dr, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Dermatology 2
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitiligo patients (Experimental)
  Interventions: Other: skin biopsy
- controls (Experimental)
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy — Lesional skin biopsy was taken from every patient. Also a skin biopsy was taken from every control subject

SUMMARY:
study & verify the hypothesis of the involvement of TSLP in the pathogenesis of vitiligo in comparison to their levels in the healthy control persons.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with generalized non-segmental vitiligo.

  * Both sexes.
  * Age < 18 years old age.
  * New cases or cases not receiving any medication for at least 3 months ago.

Exclusion Criteria:

* • Age: Patients < 18 years.

  * Segmental or universal vitiligo.
  * Pregnant and lactating females. Autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Expression levels of TSLP in patients of Vitiligo. | 7 months